CLINICAL TRIAL: NCT04788914
Title: Circulating Long Noncoding RNA as a Biomarker to Assess the Therapeutic Impact of Oral Uremic Toxin Absorbent ± Probiotics in Chronic Kidney Disease Patients With Peripheral Arterial Disease
Brief Title: lncRNAs as a Biomarker to Assess the Therapeutic Impact of Oral Absorbent ± Probiotics in CKD Patients With PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201907105MINC
Record Dates: First submitted 2020-05-19; First posted 2021-03-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: CKD; PAD
Keywords: Bamboo charcoal; LncRNA; gut microbiota; CKD; PAD; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active bamboo charcoal (Other): In this proposal, investigators aim to determine the therapeutic impact of a carbonaceous oral adsorbent made of activated bamboo charcoal (ABC) with/without probiotics on the endothelial/vascular function, CV outcome and mortality in CKD patients with PAD. In addition, investigators hypothesize that circulating long noncoding RNA (lncRNA) expression profiles and metabolome may serve as a sensitive and reliable biomarker to predict the adverse CV outcomes and death in CKD patients with established PAD. In addition, it is hypothesized that circulating lncRNAs and linked to adverse CV outcomes in CKD patients with PAD are associated with dysbiosis of gut microbiota. Investigators also hypothesize that the administration of ABC could normalize the dysbiosis of gut microbiota, dysregulated circulating lncRNAs and metabolome that are linked to adverse CV/limb outcomes in CKD patients with PAD.
  Interventions: Dietary Supplement: Active bamboo charcoal± probiotics
- Probiotics (Other): The therapeutic impact of probiotics on circulating long noncoding RNA (lncRNA) expression profiles and metabolome may serve as a sensitive and reliable biomarker to predict the adverse CV outcomes and death in CKD patients with established PAD. In addition, it is hypothesized that circulating lncRNAs and linked to adverse CV outcomes in CKD patients with PAD are associated with dysbiosis of gut microbiota.
  Interventions: Dietary Supplement: Active bamboo charcoal± probiotics

INTERVENTIONS:
Dietary Supplement: Active bamboo charcoal± probiotics — Active bamboo charcoal 2g, TID probiotics 0.8g

SUMMARY:
Participants with chronic kidney disease (CKD) are at a higher risk of developing atherosclerotic peripheral artery disease (PAD). Retention of uremic toxins such as indoxyl sulfate (IS), p-cresyl sulfate (PCS) and trimethylamine N-oxide (TMAO) during CKD is detrimental to endothelial and vascular function and can predispose to the development and progression of PAD. Many of the uremic toxins originate from gut microbial metabolism. Removal of these uremic toxins by carbonaceous oral adsorbent is beneficial, slowing down the deterioration of renal function and delaying the need for dialysis in CKD patients. However, if carbonaceous oral adsorbent could also improve vascular function and clinical outcomes in CKD patients with established PAD, remains unknown.

In this proposal, the investigators aim to determine the therapeutic impact of a carbonaceous oral adsorbent made of activated bamboo charcoal (ABC) with/without probiotics on the endothelial/vascular function, CV outcome and mortality in CKD patients with PAD. In addition, the investigators hypothesize that circulating long noncoding RNA (lncRNA) expression profiles and metabolome may serve as a sensitive and reliable biomarker to predict the adverse CV outcomes and death in CKD patients with established PAD. In addition, it is hypothesized that circulating lncRNAs and linked to adverse CV outcomes in CKD patients with PAD are associated with dysbiosis of gut microbiota. The investigators also hypothesize that the administration of ABC could normalize the dysbiosis of gut microbiota, dysregulated circulating lncRNAs and metabolome that are linked to adverse CV/limb outcomes in CKD patients with PAD.

This will be a prospective, randomized, open-labeled, blinded end-point trial for 6 months, followed by integrated assessment of endothelial/vascular function, changes in conventional athero- and inflammation-relevant biomarkers, circulating long noncoding RNAs, metabolome, and gut microbiota at baseline, ends of the 3rd and 6th month, as well as clinical CV, renal and limb outcomes up to 3 years.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-labeled, blinded end-point (so called PROBE) trial for 6 months. All patients presented to the clinics of participating sites with advanced CKD with eGFR 15 < eGFR < 60 ml/min/1.73m2 and symptomatic PAD will be screened for eligibility. The other healthy adults will be enrolled as control.

Participants who fulfill the inclusion/exclusion criteria will be invited to participate in the current study. After the participants provides the written informed consents, detailed demographic data including genders, ages, body weights, body heights, smoking status (never, past, or active), the baseline creatinine (the nadir value in the past three months) and its corresponding eGFR and CKD stages, degrees of albuminuria (Urine albumin creatinine ratio, UACR), NYHA functional class, presence of atrial fibrillation, prior cardiovascular disease (CVD, including myocardial infarct, peripheral arterial occlusive diseases), presence of diabetes mellitus (DM), or hypertension. Detailed medication list will also be obtained, with the focus on angiotensin receptor blocker or angiotensin converting enzyme inhibitors, statins, and beta-blockers.

The etiology of kidney injury will be non-mutual-exclusively categorized as:

1. Hypertensive kidney disease, participants who received any kind of anti-hypertensive drugs.
2. Diabetic kidney disease, patients who received any kind of anti-diabetics drugs.
3. Glomerulonephritis, patients who have proteinuria more than 0.5mg/dL and kidney biopsy approved Glomerulonephritis.

Eligible 120 participants (group I) with eGFR 15 < eGFR < 60 ml/min/1.73m2 and symptomatic PAD will be randomized into ABC-treatment (A) or no-treatment (B)participants with a 1:1 ratio. The other 60 eligible controls (eGFR > 60 ml/min/1.73m2 and no PAD, group II) will be also randomized into ABC-treatment (A) or no-treatment (B) with a 1:1 ratio. The participants will receive CharXenPlus 4g (with ABC 2g) thrice daily for 6 months in subgroups IA and IIA, while the participants in subgroups IB and IIB will not receive any ABC. The subgroups IA and IB will be further randomly subdivided into IAa, IAb, IBa, and IBb subsubgroups. All the participants will receive probiotics APL-MIX2 (CharXprob) 0.8 g once a day in the last 3 months except those in subsubgroups IAb and IBb.

After being processed, urine, stool, and plasma samples will be stored in -80°C for further examinations. The names and chart numbers participants will be masked to provide adequate privacy. The coding book connecting codes and individual participants will be filed separately in order to protect participants' privacy. participants will be asked if investigators can keep the encrypted samples refrigerated for 10 years for further investigations.

ELIGIBILITY:
Inclusion Criteria:

I: Patients

1. Age > 20 years old on the day of screening.
2. CKD patients with eGFR 15 < eGFR < 60 ml/min/1.73m2 in a stable status, creatinine elevated less than 0.3 mg/dL in at least 30 days before enrollment.
3. Symptomatic PAD with Rutherford Stage ≥ 2 and ABI < 0.9 (or documented by CT-angio, vascular duplex, etc.).

II: Controls

1. Age > 20 years old on the day of screening.
2. With eGFR > 60 ml/min/1.73m2
3. No clinical PAD.

Exclusion Criteria:

1. Baseline estimated glomerular filtration rates (eGFR) < 15 ml/min/1.73m2 according to MDRD equation.
2. Patients in severe malnutrition status, albumin less than 2.0 g/dL
3. Patients in severe anemia or active gastrointestinal bleeding with hemoglobulin < 8 g/dL.
4. Peptic ulcer, esophageal varices, ileus or under fasting status
5. Previous gastrointestinal operation.
6. Chronic constipation, as defined with less than 3 bowel movements per week, straining, hard stools, incomplete evacuation and inability to pass stool. If usage of oral laxatives can achieve bowel movement, this patient will not be excluded.
7. Patients with major hemorrhage, as defined with acute hemorrhage and requirement of blood transfusion during index admission.
8. Patients with a biopsy proved or clinically diagnosed advanced liver cirrhosis, Child classification B or C.
9. Solid organ or hematological transplantation recipients.
10. Patients with oliguric kidney injury, as defined with less than 500 cc/day.
11. Evidence of obstructive kidney injury or polycystic kidney disease.
12. Antibiotics or probiotics treatment within the last 2 weeks before enrollment and during follow-up period.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The change of the six-minute walk test | baseline, 3th month and 6th month
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
The change of ABI | baseline, 3th month and 6th month
  The ABI value is determined by taking the higher pressure of the 2 arteries at the ankle, divided by the brachial arterial systolic pressure.

SECONDARY OUTCOMES:
The change of InCRNA | baseline, 3th month and 6th month
  Long non-coding RNAs (long ncRNAs, lncRNA) are a type of RNA, defined as being transcripts with lengths exceeding 200 nucleotides that are not translated into protein.
The change of microbiota | baseline, 3th month and 6th month
  Gut flora
The change of EPC | baseline, 3th month and 6th month
  Circulating endothelial progenitor cells (EPCs)
The change of eGFR | baseline, 3th month and 6th month
  eGFR is estimated GFR calculated by the abbreviated MDRD equation : 186 x (Creatinine/88.4)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if black).
The change of UACR | baseline, 3th month and 6th month
  Urine albumin divided by urine creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Chau chung Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No